CLINICAL TRIAL: NCT01572857
Title: Correlation Between the Urinary Protein/Creatinine Ratio in a Single Urine Sample Versus 24-hour Proteinuria in Patients With Multiple Myeloma.
Brief Title: Urinary Protein/Creatinine Ratio in a Single Urine Sample Versus 24-hour Proteinuria in Patients With Multiple Myeloma
Acronym: RCP-MM
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201O-AOI354-35
Record Dates: First submitted 2012-03-28; First posted 2012-04-06 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; Proteinuria; Albuminuria; Urinary FLC; Urine creatinine
MeSH Terms: conditions — Multiple Myeloma; Proteinuria; Albuminuria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Proteinuria
  * Albuminuria
  * Urinary FLC (Freelite ™)
  * Urine creatinine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- first phase: This first phase aims to study the variations in urinary excretion of FLC immunoglobulin during the day and night to determine the appropriate time of day for collection of urine.
  20 patients hospitalized.
  Interventions: Biological: urinary excretion of FLC immunoglobulin
- Second phase: Determination of creatinine in 24 hours by measuring the creatinine of 24 hours 3 days in a row. This value will check the quality of urine collection for 24 hours during the study.
  30 patients hospitalized.
  Interventions: Biological: urinary excretion of FLC immunoglobulin

INTERVENTIONS:
Biological: urinary excretion of FLC immunoglobulin — First phase :
  Collection of four urine samples daily for 2 days:
  * Of the 24-hour urine
  * at 8 AM
  * at 12 AM
  * at 4 PM
  On each of these urine samples, the following analysis will be performed:
  * Proteinuria
  * Albuminuria
  * Urinary FLC (Freelite ™)
  * Urine creatinine
  Second phase:
  Determination of creatinine in 24 hours by measuring the creatinine of 24 hours 3 days in a row.
  Other Names: Non applicable.

SUMMARY:
The measurement of 24-hour proteinuria allows an assessment of treatment response in patients with multiple myeloma. But it is difficult and restrictive to make.

This study was therefore designed to investigate the correlation between the ratio of proteinuria / creatinine on samples, easier to obtain, and the 24-hour proteinuria in assessing response to this treatment .

DETAILED DESCRIPTION:
The measure of 24-hour proteinuria is an important biomarker for multiple myeloma.

Multiple myeloma is often accompanied by proteinuria overhead of secretion by plasma cells of large quantities of immunoglobulin free light chains (FLC) kappa or lambda. This proteinuria is composed of monoclonal FLC. The measure of the urinary concentration of FLC is an important biomarker for both diagnosis and evaluation of response to treatment of light chain multiple myeloma but also in intact immunoglobulins multiple myeloma.

The 24-hour proteinuria coupled with urine protein electrophoresis is the standard method for measuring the concentration of urinary FLC. However, it is difficult to obtain a reliable collection of the urine of 24 hours which can make it difficult to assess response to therapy in some patients. It would be interesting to assess proteinuria in a single urine sample collected at any time of day.

Contribution of urinary protein/creatinine ratio for assessment of proteinuria of glomerular origine.

For reasons of convenience, the extent of 24-hour proteinuria was increasingly abandoned by nephrologists in favor of urinary protein/creatinine ratio (UPCR). The use of UPCR measured on a sample of urine overcomes the inaccuracies related to the collection of 24 or variations in urine concentration. This report has been validated against the 24-hour proteinuria for screening or monitoring of renal glomerular diseases by the French Society of Nephrology. In theory, the UPCR is measured on a urine sample, taken preferably in the morning. In practice, the precision of a measurement at any time of day is quite acceptable.

Using the urinary protein/creatinine ratio for assessment of response in multiple myeloma?

The use of UPCR has been validated in patients with renal glomerular disease and especially in diabetic nephropathy. However, the UPCR has not been validated for the assessment of proteinuria overload such as those seen in myeloma. Two recent papers have studied the UPCR in multiple myeloma. The results of these articles suggest:

* That the UPCR is well correlated with the 24-hour proteinuria
* The UPCR varies over time depending on the response to treatment and could therefore be used to monitor patients on treatment

However, given their limits, these two articles do not alow to recommend the widespread use of UPCR instead of the classic 24-hour proteinuria in clinical practice yet. Prospective studies are needed to analyze the correlation between UPCR and proteinuria of 24 hours to assess response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* For the first part of the study :

  * adult patient
  * giving a free, informed and written consent
  * patient having a follow-up in the service for multiple myeloma, whatever the age of diagnosis, the isotype of monoclonal component, stage and disease activity
  * patient hospitalized in the service whatever the reason for hospitalization (related or not with multiple myeloma)
  * proteinuria ≥ 500 mg/24h
  * percentage of albuminuria < 50% on urinary protein electrophoresis
  * presence of immunoglobulin FLC in immunofixation of urine proteins
* For the second part of the study :

  * adult patient
  * giving a free, informed and written consent
  * patient having a follow-up in the service for multiple myeloma, whatever the age of diagnosis, the isotype of monoclonal component
  * requiring the initiation of treatment with chemotherapy
  * proteinuria ≥ 500 mg/24h
  * percentage of albuminuria < 50% on urinary protein electrophoresis
  * presence of immunoglobulin FLC in urine proteins immunofixation

Exclusion Criteria:

* minor patient
* proteinuria < 500 mg/24h
* predominantly glomerular proteinuria with ≥ 50% albumin on urinary protein electrophoresis
* absence of immunoglobulin FLC in urine proteins immunofixation
* progressive urinary infection
* patient with a glomerular nephropathy
* macroscopic hematuria
* patient unable to perform a urinary collection for 24 hours
* patient unable to give a consent
* pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple myeloma.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2018-01 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
change in urinary protein/creatinine ratio | Change from baseline in urinary protein/creatinine ratio at 8 AM, 12 AM, 4 PM
  To study the correlation between the urinary protein/creatinine ratio in the sample and 24-hour proteinuria in the assessment of treatment response in patients with multiple myeloma.

SECONDARY OUTCOMES:
changes in urinary excretion of FLC | Of the 24-hour urine, at 8 AM, 12 AM, 4 PM
  To study the changes in urinary excretion of FLC during the day and night
methods for estimating the urinary concentration of FLC | Of the 24-hour urine, at 8 AM, 12 AM, 4 PM
  Compare different methods for estimating the urinary concentration of FLC

CONTACTS AND LOCATIONS:
Overall Officials: Olivier DECAUX, MD, Principal Investigator — Service de Medecine interne - Hôpital Sud - Rennes
Locations (1):
- Service de Médecine interne - Hôpital Sud : Rennes University Hospital, Rennes, France